CLINICAL TRIAL: NCT06390878
Title: Nationwide Research on the Rewilding of Kindergarten Yards - Vahvistu
Brief Title: Nationwide Research on the Rewilding of Kindergarten Yards
Acronym: Vahvistu
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Resources Institute Finland (Other Government)
Collaborators: Tampere University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R24023
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Microbial Colonization; Atopic Dermatitis; Asthma in Children; Allergy; Cognitive Change; Respiratory Infection; Nature, Human
Keywords: Commensal microbiome; Atopy; Planetary health; Biodiversity; Cognitive skills
MeSH Terms: conditions — Communicable Diseases; Dermatitis, Atopic; Hypersensitivity; Respiratory Tract Infections | interventions — Biodiversity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rewilding (Experimental): The kindergarten yards are modified with natural elements to increase children's exposure to biodiversity and playground equipment are incorporated to the yards to increase children's physical activity.
  Interventions: Other: Biodiversity
- Control (Experimental): The kindergarten yards are not rewilded with natural elements and the biodiversity is low at the yards. Playground equipment are incorporated to the yards to increase children's physical activity.
  Interventions: Other: Playground equipment

INTERVENTIONS:
Other: Biodiversity — In rewilding kindergartens, the yards are modified with biological elements, i.e., vegetation and plantation will be added to the yards.
  Arms: Rewilding
Other: Playground equipment — Playground equipment that increase the physical activity of children will be added to the kindergarten yards.
  Arms: Control

SUMMARY:
Biodiversity is essential for nature and human well-being. Land use has reduced biodiversity in cities that is associated with altered commensal microbiota and a rising burden of immunological disorders among urban children.

The investigators will estimate how rewilding of kindergarten yards affects commensal microbiome, prevalence of allergies, asthma, atopic dermatitis and infections, cortisol levels, cognitive skills and plasma cytokine levels of children.

Our specific aims are:

To assess if rewilding diversifies health-associated skin, saliva and gut microbiota and reduces infectious diseases and atopic or allergic symptoms.

Assess whether the rewilding has positive effects on cognitive skills. Assess whether the rewilding changes cortisol and plasma cytokine levels. The investigators will recruit altogether 320 (160 per treatment) study subjects aged between 1-5 to questionnaire study (Task 2), from which 120 study subjects will be analyzed more detailed using microbiological and blood samples (Task 1).

ELIGIBILITY:
Inclusion Criteria:

* Attendance in kindergarten

Exclusion Criteria:

* Use of antibiotics in the year before sampling

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Skin Gammaproteobacteria | Baseline, 3 month, 1 year, 2 year, 3 year
  Difference on skin gammaproteobacterial diversity between rewilding and control group

SECONDARY OUTCOMES:
Cortisol levels | Baseline, 3 month, 1 year, 2 year, 3 year
  Cortisol levels measured from hair samples
Difference in diversity of skin, saliva and stool microbiota | Baseline, 3 month, 1 year, 2 year, 3 year
  It will be analyzed if microbial communities are different between treatments
Microbial observed species richness | Baseline, 3 month, 1 year, 2 year, 3 year
  Higher score in observed species richness of commensal microbiota among biodiversity treatment
Difference in taxonomies of skin, saliva and stool microbiota | Baseline, 3 month, 1 year, 2 year, 3 year
  It will be analyzed if microbial communities are different between treatments
White blood cell distribution | Baseline, 3 month, 1 year, 2 year, 3 year
  It will be analyzed if the distribution is different between treatments
White blood cell transcriptomics | Baseline, 3 month, 1 year, 2 year, 3 year
  White blood cell transcriptome is analyzed with single cell RNA sequencing.
Plasma cytokines | Baseline, 3 month, 1 year, 2 year, 3 year
  Cytokines will be analyzed analyzed with Meso Scale.
Skin cytokines | Baseline, 3 month, 1 year, 2 year, 3 year
  Cytokines will be analyzed using skin tape strip samples.
Infectious diseases | Baseline, 3 month, 1 year, 2 year, 3 year
  Infections will be recorded with questionnaires.
Asthma symptoms | Baseline, 3 month, 1 year, 2 year, 3 year
  Asthma symptoms will be recorded with questionnaires.
Atopic dermatitis | Baseline, 3 month, 1 year, 2 year, 3 year
  Atopic dermatitis will be recorded with questionnaires.
Allergy | Baseline, 3 month, 1 year, 2 year, 3 year
  Allergies will be recorded with questionnaires.
Patient-oriented Eczema Measure | Baseline, 3 month, 1 year, 2 year, 3 year
  Lower score on patient-oriented Eczema Measure among intervention treatment compared to control that indicates lower eczema among intervention treatment. Minimum 0, maximum 28.
Wechsler Preschool and Primary Scale of Intelligence | Baseline, 3 month, 1 year, 2 year, 3 year
  Higher score on Wechsler Preschool and Primary Scale of Intelligence among intervention treatment compared to control that indicates better cognitive skills among intervention treatment. Minimum 40, maximum 170.

OTHER OUTCOMES:
Associations between environmental factors and cytokine levels. | Baseline, 3 month, 1 year, 2 year, 3 year
  It will be analyzed if environmental factors correlate with cytokine levels.
Associations between environmental factors and commensal microbiota. | Baseline, 3 month, 1 year, 2 year, 3 year
  It will be analyzed if environmental factors correlate with richness of commensal microbiota.
Associations between environmental factors and white blood cells | Baseline, 3 month, 1 year, 2 year, 3 year
  It will be analyzed if environmental factors correlate with white blood cell distributions.
Associations between environmental factors and cortisol levels | Baseline, 3 month, 1 year, 2 year, 3 year
  It will be analyzed if environmental factors correlate with cortisol levels.
Associations between environmental factors and cognitive skills. | Baseline, 3 month, 1 year, 2 year, 3 year
  It will be analyzed if environmental factors correlate with cognitive skills.
Associations between environmental factors and infectious diseases. | Baseline, 3 month, 1 year, 2 year, 3 year
  It will be analyzed if environmental factors correlate with the prevalence of infectious diseases.
Associations between environmental factors and atopy. | Baseline, 3 month, 1 year, 2 year, 3 year
  It will be analyzed if environmental factors correlate with the atopic dermatitis
Associations between environmental factors and allergies. | Baseline, 3 month, 1 year, 2 year, 3 year
  It will be analyzed if environmental factors correlate with the allergy symptoms.
Associations between environmental factors and asthma. | Baseline, 3 month, 1 year, 2 year, 3 year
  It will be analyzed if environmental factors correlate with the asthma symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Aki Sinkkonen, Principal Investigator — Natural Resources Institute Finland
Locations (2):
- Finland (2):
  - Natural Resources Institute Finland, Helsinki, Uusimaa
  - Tampere University, Tampere